CLINICAL TRIAL: NCT06891898
Title: iLet Dosing Decision Software Postmarket Surveillance Plan (PS240001): The iLet Experience Study
Brief Title: The iLet Experience Study
Status: Recruiting | Type: Observational
Sponsor: Beta Bionics, Inc. (Industry)
Collaborators: The Scripps Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PS240001
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; postmarket registry; iLet Bionic Pancreas; Beta Bionics; iLet Dosing Decision Software
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: No

GROUPS / COHORTS (1):
- iLet Bionic Pancreas: users of the iLet Bionic Pancreas installed with the iLet Dosing Decision Software
  Interventions: Device: iLet Dosing Decision Software

INTERVENTIONS:
Device: iLet Dosing Decision Software — Interoperable alternate glycemic controller
  Other Names: iLet Bionic Pancreas

SUMMARY:
A one-year, prospective single-arm cohort study to collect safety and effectiveness data on the iLet Dosing Decision Software during real-world use in people 6 years of age or older with type 1 diabetes (T1D) with 12 months follow-up.

DETAILED DESCRIPTION:
The study will compare outcomes data during iLet use to efficacy and safety outcomes data derived from epidemiological studies, such as data published by the T1D Exchange registry, and to the results of the Bionic Pancreas Pivotal Trial (BPPT), with a special emphasis on serious adverse effects such as severe hypoglycemia and DKA. An analysis will be conducted comparing glycemic outcomes during iLet use to baseline pre-iLet CGM and HbA1c data in participants who have provided this data. In addition, the study will determine the frequency and types of anticipated and unanticipated device issues experienced by users during real-world use.

ELIGIBILITY:
Inclusion Criteria:

* Users must meet the following criteria in order to be enrolled in the study:

  1. Diagnosed with type 1 diabetes and prescribed the iLet Bionic Pancreas System
  2. At least 6 years of age
  3. Using or planning to use either U100 Novolog (insulin aspart) or U100 Humalog (insulin lispro) in ready-to-fill cartridges, or U100 Fiasp® PumpCart® (insulin aspart) in pre-filled 1.6mL cartridges
  4. Willing to provide HbA1c results obtained within the 6-month period prior to starting use of the iLet and during the last 6-months of study participation
  5. Willing to provide CGM data, if available, obtained in the 1-month period prior to starting use of the iLet
  6. For females, not pregnant or planning pregnancy in the next 12 months
  7. Able to respond to alerts and alarms, and to provide basic diabetes self-management
  8. Reside full-time in the US
  9. Able to speak and read English
  10. Willing and able to download the iLet Mobile App and keep it active throughout the study and upload device data regularly
  11. Willing to answer baseline survey, monthly surveys, and share CGM data, and follow-up data, as necessary

Exclusion Criteria:

* Users with the following characteristics will not be considered candidates for the study:

  1. Type 2 diabetes, cystic fibrosis-related diabetes, congenital hyperinsulinism, pancreatogenic diabetes, or any form of diabetes mellitus other than type 1 diabetes
  2. Use or planned use of any insulin in the iLet other than U100 Novolog (insulin aspart) or U100 Humalog (insulin lispro) in ready-to-fill cartridges, or U100 Fiasp® PumpCart® (insulin aspart) in pre-filled 1.6mL cartridges
  3. End-stage renal disease on renal replacement therapy (peritoneal dialysis or hemodialysis)
  4. Use or planned use of hydroxyurea

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will include users of the iLet Dosing Decision Software who are at least 6 years old and have been diagnosed with Type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 1875 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Severe Hypoglycemia/cognitive impairment | 1 year
  Number of severe hypoglycemia events associated with cognitive impairment requiring the assistance of a third party for treatment per 100 patient years

SECONDARY OUTCOMES:
Severe Hypoglycema/unconsciousness or seizure | 1 year
  Number of severe hypoglycemia events associated with unconsciousness or seizure per 100 patient years
DKA | 1 year
  Number of diabetic ketoacidosis events per 100 patient years
Unanticipated Adverse Device Effects | 1 year
  Rate of unanticipated adverse device effects
Mean CGM Glucose | 1 year
  Mean glucose as determined by CGM after 1 year of iLet use
Time < 54 mg/dL | 1 year
  Percentage of time with CGM glucose < 54 mg/dL
Time < 70 mg/dL | 1 year
  Percentage of time with CGM glucose < 70 mg/dL
Time in Range | 1 year
  Percentage of time with CGM glucose 70-180 mg/dL
Time > 180 mg/dL | 1 year
  Percentage of time with CGM glucose > 180 mg/dL
Time > 250 mg/dL | 1 year
  Percentage of time with CGM glucose > 250 mg/dL
Rate of CGM-determined hypoglycemic events | 1 year
  Rate of hypoglycemic events defined as at least 15 consecutive minutes of CGM glucose < 54 mg/dL - the hypoglycemic event ends when there are at least 15 consecutive minutes with a CGM glucose greater than or equal to 70 mg/dL and the participant becomes eligible for another hypoglycemic event
Rate of CGM-determined hyperglycemic events | 1 year
  Rate of hyperglycemic events defined as at least 90 cumulative minutes with a CGM glucose value > 300 mg/dL within a 120-minute period - the hyperglycemic event ends when there are at least 15 consecutive minutes with a CGM glucose value less than or equal to 180 mg/dL and the participant becomes eligible for another hyperglycemic event.
Mean glucose coefficient of variation | 1 year
  Mean CGM glucose Intrasubject coefficient of variation
Time in BG-Run mode | 1 year
  Percent of time spent in BG-run mode
Time in BG-run mode for longer than 4 hours | 1 year
  Percent of time spent in BG-run mode episodes longer than 4 hours
Severe Hypoglycemia During BG-run mode | 1 year
  Rate of severe hypoglycemic events beginning during a BG-run mode episode that lasted more than 4 hours or within 6 hours of a BG-run episode that lasted more than 4 hours
DKA During BG-run mode | 1 year
  Rate of diabetic ketoacidosis events during a BG-run mode episode that lasted more than 4 hours or within 6 hours of a BG-run episode that lasted more than 4 hours
Unanticipated Adverse Device Effects during BG-run mode | 1 year
  Rate of unanticipated adverse device effects during BG-run mode
Average duration of BG-run mode episodes | 1 year
  Average duration of BG-run mode episodes
Percentage of time insulin suspended during BG-Run episodes >4 hours | 1 year
  During BG-run mode episodes that lasted more than 4 hours, percentage of time no insulin could be delivered as a result of failure to enter BG values at the required intervals
Mean CGM glucose at time of entry into BG-run episodes >4 hours | 1 year
  Mean CGM glucose at the time of entry into BG-run mode episodes that lasted more than 4 hours
Mean CGM glucose at time of exit from BG-run episodes >4 hours | 1 year
  Mean CGM glucose at the time of exit from BG-run mode into CGM-run mode after episodes of BG-run mode that lasted more than 4 hours
Insulin TDD | 1 year
  Insulin total daily dose (u/kg/day)
Mean Baseline HbA1c of all Participants | Baseline
  The last available baseline HbA1c value (when available) will be reported as the mean ± standard deviation.
Mean HbA1c on iLet | 1 year or final available during study period
  The last available HbA1c value during the study period (when available) will be reported as the mean ± standard deviation.
Mean change in HbA1c | 1 year or final available during study period compared to baseline
  The change in HbA1c from the last available baseline value to the last available value during the study period (when both values are available) will be reported as the mean ± standard deviation.

OTHER OUTCOMES:
Mean number of swipes to unlock the iLet per day | 1 year
  Mean number of swipes to unlock the iLet per day
Mean number of total meal announcements made per day | 1 year
  Mean number of meal announcements made per day - total regardless of meal type
Average number of breakfast announcements made per day | 1 year
  Mean number of total breakfast announcements made per day
Average number of lunch announcements made per day | 1 year
  Mean number of total lunch announcements made per day
Average number of dinner announcements made per day | 1 year
  Mean number of total dinner announcements made per day

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Beta Bionics
Locations (1):
- Beta Bionics, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
It has not yet been decided if IPD will be shared.